CLINICAL TRIAL: NCT01005758
Title: DFCI ALL Adult Consortium Protocol: Adult ALL Trial
Brief Title: Combination Chemotherapy in Treating Adult Patients With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: William G. Blum, Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000632144; OSU-08066; 2008C0112; DFCI-06254
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-10

CONDITIONS: Leukemia
Keywords: untreated adult acute lymphoblastic leukemia; Philadelphia chromosome positive adult precursor acute lymphoblastic leukemia; L1 adult acute lymphoblastic leukemia; L2 adult acute lymphoblastic leukemia; T-cell adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; etoposide phosphate; Hydrocortisone; Imatinib Mesylate; Mercaptopurine; Methotrexate; Methylprednisolone; pegaspargase; Prednisolone; Prednisone; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: cytarabine
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: etoposide phosphate
Drug: hydrocortisone sodium succinate
Drug: imatinib mesylate
Drug: mercaptopurine
Drug: methotrexate
Drug: methylprednisolone
Drug: pegaspargase
Drug: prednisolone
Drug: prednisone
Drug: vincristine sulfate
Other: laboratory biomarker analysis
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects of combination chemotherapy and to see how well it works in treating adult patients with newly diagnosed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the feasibility, toxicity, and efficacy of a high-risk pediatric treatment regimen in adult patients with newly diagnosed acute lymphoblastic leukemia (ALL).
* To explore the relative toxicity of pegaspargase IV.
* To explore the relative efficacy and toxicity of adding imatinib mesylate to multi-agent chemotherapy for patients with Philadelphia chromosome-positive ALL.

Secondary

* To estimate the complete remission (CR) rate at the end of induction therapy and calculate the corresponding 90% confidence interval (CI).
* To estimate the disease-free survival (DFS), defined as the time from achieving a CR to the first disease recurrence or death, of a subset of patients who achieve a CR at the end of induction therapy.
* To estimate the overall survival (OS), defined as the time from study entry to death from any cause, of all patients.
* To calculate the median, 2-year, and 3-year DFS and OS rates and their corresponding 95% CI's.
* To evaluate the prognostic significance of the prednisone prophase response, minimal residual disease at various time points, the frequency and type of tyrosine kinase mutations, and gene expression profiles at diagnosis.

OUTLINE: This is a multicenter study.

* Steroid prophase therapy (for patients who have not received steroids within the past 7 days): Patients receive cytarabine intrathecally (IT) on day 0 or 1 and methylprednisolone IV 3 times daily on days 1-3.
* Induction therapy (weeks 1-4): Patients receive vincristine sulfate IV on days 4, 11, 18, and 25; doxorubicin hydrochloride IV on days 4 and 5; methotrexate IV on day 6; pegaspargase IV over 1 hour on day 7; and prednisone or prednisolone orally 2-3 times daily or methylprednisolone IV 3 times daily on days 4-32. Patients also receive methotrexate, cytarabine, and hydrocortisone IT on day 18 and methotrexate IT on day 32. After completion of induction therapy, patients with documented complete remission (CR) proceed to consolidation IA therapy (group A). Patients with partial remission proceed to consolidation IC therapy (group B). Patients with refractory disease are removed from the study.
* Consolidation I therapy (weeks 5-13): Patients are assigned to 1 of 2 groups according to their CR status.

  * Group A (patients who achieved CR by day 32 or patients with delayed recovery):

    * Consolidation IA therapy (weeks 5-7): Patients receive vincristine sulfate IV, doxorubicin hydrochloride IV, methotrexate IT, and high-dose methotrexate IV on day 1. Patients also receive oral mercaptopurine once daily on days 1-14. Patients then proceed to consolidation IB therapy.
    * Consolidation IB therapy (weeks 8-10): Patients receive cyclophosphamide IV over 1 hour and methotrexate IT on day 1, low-dose cytarabine IV or subcutaneously (SC) on days 2-5 and 9-12, and oral mercaptopurine once daily on days 1-14. Patients then proceed to consolidation IC therapy.
    * Consolidation IC therapy (weeks 11-13): Patients receive high-dose cytarabine IV over 3 hours twice daily on days 1 and 2, etoposide phosphate IV over 2 hours on days 3-5, and oral dexamethasone twice daily on days 1-5. Patients also receive pegaspargase IV over 1 hour every 2 weeks beginning on day 8 and continuing during CNS therapy and consolidation II therapy until a total of 15 doses are administered. After completion of consolidation IC therapy, patients proceed to CNS therapy.
  * Group B (patients who failed to enter a CR after 32 days of multi-agent induction chemotherapy):

    * Consolidation IC therapy (weeks 5-7): Patients receive high-dose cytarabine IV over 3 hours twice daily on days 1 and 2, etoposide phosphate IV over 2 hours on days 3-5, and oral dexamethasone twice daily on days 1-5. Patients who achieve CR at the end of consolidation IC therapy proceed to consolidation IA therapy. Patients with > 5% blast count at the end of consolidation IC therapy are removed from the study.
    * Consolidation IA therapy (weeks 8-10): Patients receive vincristine sulfate IV, doxorubicin hydrochloride IV, methotrexate IT, and high-dose methotrexate IV on day 1. Patients also receive oral mercaptopurine once daily on days 1-14. Patients then proceed to consolidation IB therapy.
    * Consolidation IB therapy (weeks 11-13): Patients receive cyclophosphamide IV over 1 hour and methotrexate IT on day 1, low-dose cytarabine IV or SC on days 2-5 and 9-12, and oral mercaptopurine once daily on days 1-14. Patients also receive pegaspargase IV over 1 hour every 2 weeks beginning on day 8 and continuing during CNS therapy and consolidation II therapy until a total of 15 doses are administered. After completion of consolidation IB therapy, patients proceed to CNS therapy.
* CNS therapy (weeks 14-16): Patients receive vincristine sulfate IV and doxorubicin hydrochloride IV on day 1, oral mercaptopurine once daily on days 1-14, oral dexamethasone twice daily on days 1-5, and pegaspargase as described in consolidation I therapy. Patients also receive methotrexate, cytarabine, and hydrocortisone IT twice weekly for 4 doses and undergo cranial irradiation once daily for 8-10 days. After completion of CNS therapy, patients proceed to consolidation II therapy.
* Consolidation II therapy (weeks 17-43): Patients receive vincristine sulfate IV and doxorubicin hydrochloride IV on day 1, oral mercaptopurine once daily on days 1-14, oral dexamethasone twice daily on days 1-5, and pegaspargase as described in consolidation I therapy. Treatment repeats every 3 weeks until patients have received a cumulative dosage of 300 mg/m^2 of doxorubicin hydrochloride and 30 post-remission weeks of pegaspargase have been administered. When patients complete doxorubicin hydrochloride, they receive methotrexate IV once weekly (except on the week that they receive methotrexate IT). Patients also receive methotrexate, cytarabine, and hydrocortisone IT every 18 weeks (first dose is given 18 weeks after the first lumbar puncture administered during CNS therapy). After completion of consolidation II therapy, patients proceed to continuation therapy.
* Continuation therapy (weeks 44-113): Patients receive vincristine sulfate IV on day 1; methotrexate IV on days 1, 8, and 15; oral mercaptopurine once daily on days 1-14; and oral dexamethasone twice daily on days 1-5. Treatment repeats every 3 weeks for a total of 104 weeks (24 months) of continued CR. Patients also receive methotrexate, cytarabine, and hydrocortisone IT every 18 weeks. Patients do not receive methotrexate IV on the week that they receive methotrexate IT.

Patients with Philadelphia chromosome-positive disease or with bcr-abl translocation on molecular studies also receive oral imatinib mesylate once daily beginning on day 14 of induction therapy and continuing until completion of continuation therapy. These patients should proceed to allogeneic stem cell transplantation as soon as feasible based on donor availability and the patient's medical status.

Bone marrow, peripheral blood, and other samples are collected periodically for research studies (including minimal residual disease analysis, gene expression profiling, and tyrosine kinase sequencing).

After completion of study treatment, patients are followed up monthly for 6 months, every 2 months for 6 months, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphoblastic leukemia (ALL)
* No known mature B-cell ALL*, defined by the presence of surface immunoglobulin, L3 morphology, t(8;14)(q24;q32), t(8;22), or t(2;8)

  * Patients with T-cell surface markers and t(8;14)(q24;q11) are eligible NOTE: *Patients with mature B-cell ALL will be removed from the study as soon as that diagnosis is made.
* No secondary ALL (i.e., ALL arising after another malignancy)

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known HIV positivity (HIV testing is not required)
* No comorbid medical condition that would, in the investigator's opinion, make participation in this study and adherence to the study guidelines a compromise to the study objectives
* No active psychiatric or mental illness that would make giving informed consent or careful clinical follow-up unlikely

PRIOR CONCURRENT THERAPY:

* No prior anti-leukemic therapy except ≤ 1 week of steroids, emergent radiotherapy to the mediastinum, hydroxyurea, or emergent leukapheresis

  * Patients who have received steroids within the past 7 days are eligible but will not receive steroid prophase therapy on study
* No concurrent chronic steroids or anti-metabolite therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-01; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intensification therapy, measured as the percentage of patients who, having achieved a complete remission after induction therapy, receive > 25 weeks of pegaspargase IV as part of intensification therapy
Toxicity

SECONDARY OUTCOMES:
Complete remission rate
Disease-free and overall survival
Prognostic significance of prednisone prophase response, minimal residual disease at various time points, tyrosine kinase mutations, and gene expression profiles at diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: William G. Blum, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center